CLINICAL TRIAL: NCT01101295
Title: The ITP-RITUX Cohort: An Observational Study on Rituximab Off-label Use for Immune ThrombocytoPenia.
Brief Title: The ITP-RITUX Cohort: Rituximab in Immune ThrombocytoPenia.
Acronym: ITP-RITUX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Khellaf Mehdi, Medical Doctor, Henri Mondor University Hospital
Other Study IDs: GECAI
Record Dates: First submitted 2010-04-05; First posted 2010-04-09 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Autoimmune Thrombocytopenia
Keywords: Immune Thrombocytopenia; Rituximab; side effects; tolerance; safety; splenectomy; serum sickness
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Serum Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of the study is to describe by a prospective observational study the serious adverse events occurring in patients treated off-label by rituximab for Immune Thrombocytopenia.

DETAILED DESCRIPTION:
Rituximab (RTX) is used in the treatment of malignant non-Hodgkin's indication for which it has been authorized since 1997 and why it is considered effective and well tolerated. Rituximab is also effective and well tolerated in combination with methotrexate in severe rheumatoid arthritis (RA) refractory to anti-TNF. To date, the RA is the only autoimmune disease in which rituximab has proven efficacy in randomized trials and has obtained authorization in this indication. There are also data from the literature, for the benefit of rituximab in other autoimmune diseases like Lupus, cryoglobulinemia associated to Hepatitis C or Sjogren's disease.

Immune Thrombocytopenia (ITP) is an autoimmune disease in which there is thrombocytopenia due in part to destruction of platelets by autoantibodies. In adults, the disease is most often chronic and in the most severe forms, the treatment of choice is splenectomy. Rituximab was suggested during chronic ITP when used with 4 weekly infusions of 375 mg/m2, 60% of patients achieve an immediate response and 30 to 40% a prolonged response. These encouraging results and the apparent good tolerance advocate for using rituximab as first-line treatment for patients refractory to splenectomy. In France, Afssaps - French Health Products Safety Agency has recently issued a temporary protocol processing to authorize rituximab in this indication. Nevertheless, many questions remain unresolved, including the tolerance of long-term treatment and the risk of late relapse in responders. This justifies the creation of this register, whose establishment is recommended by Afssaps - French Health Products Safety Agency.

ELIGIBILITY:
Inclusion Criteria:

* ITP diagnosis according to the American Society of Hematology society
* Secondary ITP if the underlying disease is an autoimmune disease(Lupus,Sjogren..)

Exclusion Criteria:

* Previous treatment by rituximab
* Secondary ITP associated to a hematologic disease (Chronic Lymphocytic Leukemia, Hodgkin Disease...)
* Secondary ITP associated to a chronic infectious disease (Hepatitis B, C, HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immune ThrombocytoPenia (ITP) patients according to the American Society of Hematology (ASH).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a serious adverse events (clinical or biological events) | 5 years
  reaction during perfusions, hypogammaglobulinemia, neutropenia,etc...

SECONDARY OUTCOMES:
Impact of rituximab on the natural history of ITP | 5 years
  Number of patients in complete response (platelet count>100G/L), in partial response (platelet count>50G/L and at least doubling the baseline platelet count)or in failure. Rate of diminution for the concomittant therapies for ITP.
  Use of emergencies treatment for ITP.
Modality of the administration of rituximab | 5 years
  number of perfusions, dosage, retreatment.
Characteristics of the patients receiving Rituximab | 5 years
  age, sex, duration of ITP, previous used treatment
Evaluation of the Platelet count evolution | 5 years
  Platelet count estimated at Month 1, 3 and then every 6 months during the 5 years of follow-up.
Rate of splenectomy in the cohort | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand GODEAU, MD, Principal Investigator — National Reference Center for Study of Cytopenia
Locations (2):
- France (2):
  - Henri Mondor University Hospital, Créteil, Val de Marne
  - National Reference Center for the Study of Auto Immune Cytopenia, Créteil, Val de Marne

REFERENCES:
- [Derived] Khellaf M, Charles-Nelson A, Fain O, Terriou L, Viallard JF, Cheze S, Graveleau J, Slama B, Audia S, Ebbo M, Le Guenno G, Cliquennois M, Salles G, Bonmati C, Teillet F, Galicier L, Hot A, Lambotte O, Lefrere F, Sacko S, Kengue DK, Bierling P, Roudot-Thoraval F, Michel M, Godeau B. Safety and efficacy of rituximab in adult immune thrombocytopenia: results from a prospective registry including 248 patients. Blood. 2014 Nov 20;124(22):3228-36. doi: 10.1182/blood-2014-06-582346. Epub 2014 Oct 7. PMID 25293768